CLINICAL TRIAL: NCT00696306
Title: Diffusion Tensor Imaging (DTI) and Susceptibility Weighted Imaging (SWI) as a Predictor of Functional Outcome in Acute Ischemic Stroke
Brief Title: MRI-SWI as a Predictor of Functional Outcome in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Chin-I Chen, MD, PhD, Taipei Medical University-Wan Fang Hospital
Other Study IDs: 2007WFCRC-002
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Acute Ischemic Stroke; Stroke; Cerebral Stroke; Cerebrovascular Accident
Keywords: Acute Ischemic Stroke; Stroke; MRI; DTI; Diffusion Tensor Imaging; SWI; Susceptibility Weighted Imaging; Outcome; Axonal Injury
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to use diffusion tensor imaging (DTI) derived axial diffusivity and susceptibility weighted imaging (SWI) to evaluate the severity of acute ischemic stroke and to predict its functional outcome.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death in Taiwan. The morbidity and mortality of stroke is also very high worldwide. In the United States, about one third of 800,000 stoke patients became disabled; while in Taiwan, 13,000 out of 68,000 stroke patients died each year.

Diffusion tensor imaging (DTI) characterizes the three-dimensional distribution of water diffusion, which is highly anisotropic. Previous studies utilized DTI derived mean diffusivity (MD) and fractional anisotropy (FA) have found correlation between pathological changes of white matter and prognosis of stroke. However, the result was not specific due to the reason that any change at either axon or myelin sheath resulted in FA reduction. DTI, on the other hand, differentiate morphological change at axon and myelin sheath with axial and radial diffusivity, respectively. With this data, we hypothesized that the prognosis might be more relevant to pathological change with axon post-stroke when compare to Diffusion-Weighted imaging (DWI)/Apparent Diffusion Coefficient (ADC).

Susceptibility-weighted imaging (SWI) is a newer technique which use fully velocity compensation gradient echo sequence to receive magnitude and phase imaging. SWI can be used to detect early phase bleed, intra-arterial thrombus, cerebral venous thrombosis, thus evaluate the prognosis of patients by detect leptomeningeal collateral circulation and intravascular deoxygenation changes. We hypothesized that the prognosis is better in post-stroke patients with preserved leptomeningeal collateral circulation and venous circulation of large blood vessel. Therefore, we conduct the study to use DTI derived axial diffusivity and SWI to evaluate the severity and to predict the functional outcome in acute ischemic stroke patient.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 20 years
* Patients with acute pathological changes in CNS within 7 days admitted from outpatient, ER, or inpatient department
* Confirmed diagnosis of acute ischemic stroke by clinical testings and CT scan performed by a neurologist
* Signed informed consent from patient

Exclusion Criteria:

* Any person with pacemaker, metal implant, claustrophobia, or any other contraindication for MR examination
* Any person with epilepsy, brain hematomas, brain tumor, or any neurological disease confirmed by CT scan
* Any other clinical condition which, in the opinion of the principal investigator, would not be suitable for this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Ischemic Stroke
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To correlate the prognosis of acute ischemic stroke with the result of MRI-DTI and the result of SWI. | 6 months

SECONDARY OUTCOMES:
To establish the DTI/SWI protocol as the biomarker for future research in neurological disorders, such as brain tumor, brain injury, brain developmental disorders, and Multiple Sclerosis. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chin-I Chen, MD, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan